CLINICAL TRIAL: NCT03590041
Title: Invested in Diabetes: Comparing Patient-Centered Outcomes of Standardized Versus Patient-Driven Diabetes Shared Medical Appointments (PCORI IHS-1609-36322)
Brief Title: Comparative Effectiveness of Diabetes Shared Medical Appointment Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-2377
Record Dates: First submitted 2018-06-15; First posted 2018-07-18 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus Type 2, Comparative Effectiveness Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The two interventions are based in the Chronic Care Model, which emphasizes whole person care, addressing physical, mental health and psychosocial needs. The conceptual model underlying patient-driven diabetes Shared Medical Appointments is based on self-determination theory (SDT) and principles of whole person care. According to SDT, human motivation and behavior are a function of the social environment and the extent to which that environment supports basic psychological needs shown to enhance "self-determined motivation."
Masking Description: Blinding is not possible with the study design. Patients will not know that there is a difference in SMAs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized SMA (Active Comparator): The standardized SMA model includes the same TTIM curriculum as in the patient-driven model, but it is delivered in a standardized way (order of and time spent on topics are set) across all participating practices.
  Interventions: Behavioral: Standardized SMA
- Patient-driven SMA (Active Comparator): In the patient-driven SMA model, patients receive the same TTIM curriculum, but patients at each practice are able to set the order of the curriculum and dictate how long to spend on each topic.
  Interventions: Behavioral: Patient-driven SMA

INTERVENTIONS:
Behavioral: Standardized SMA — Patients receiving the Standardized SMA intervention will be part of group visits that cover a modified TTIM 6-session curriculum, delivered only by health educators. The Standardized SMA approach will be uniformly administered at each practice. Topics will be covered in a predetermined order and patients will not have a say in terms of what content they wish to cover. Patients receive the Standardized SMA approach if their practice is randomly assigned to the Standardized SMA arm. Practices are cluster-randomized to deliver a standardized or patient-driven group visit model.
  Arms: Standardized SMA
Behavioral: Patient-driven SMA — Patients receiving the Patient-driven SMA intervention will be part of group visits that cover a modified TTIM 6-session curriculum, but patients are in control of time spent and order of the topics. The Patient-driven SMA will be delivered by a multidisciplinary team consisting of a Health Educator, medical provider, Behavioral Health Professional, and a diabetes peer mentor. Patient-driven SMAs may be delivered differently at each practice, as patients choose the topics that are most important to spend the most time on. All topics will be covered, but the order and time spent is up to the group. Patients receive the Patient-driven SMA approach if their practice is randomly assigned to that arm. Practices are cluster-randomized to deliver a standardized or patient-driven SMA model.
  Arms: Patient-driven SMA

SUMMARY:
In this study, the investigators will compare the effectiveness of patient-driven diabetes Shared Medical Appointments (SMAs) to standardized diabetes SMAs. The curriculum to be used is Targeted Training for Illness Management (TTIM), a 6-session modular group intervention for chronic illness self-management, and has been tested in diabetes. The standardized group visit model will consist of diabetes SMAs with the full TTIM 6-session curriculum, led by a health educator.

DETAILED DESCRIPTION:
Type II Diabetes is a prevalent chronic disease with poor outcomes, and requires daily self-care, including blood glucose monitoring, following a diabetes-friendly diet, engaging in regular physical activity, and medication adherence. Patients with diabetes benefit from comprehensive diabetes self-management education (DSME) and self-management support (SMS) in primary care. Shared medical appointments (SMAs) are one way to efficiently and effectively provide DSME and SMS. SMAs can have a variety of different features, but it is not known which features are most effective for which types of patients. Patients and other stakeholders engaged in planning this study proposed a model with "diabetes' veterans" (i.e., diabetes peer mentors) who co-facilitating group visits with a variety of diabetes care professionals, and then working one-on-one with patients to help apply what they learned. The group visit curriculum should include topics on physical activity, healthy eating, taking medication, acceptance and coping, and social support, and each cohort of patients should get to select topics most relevant to them. The practice stakeholders want to do more comprehensive group visit models, but need to know the extent to which SMA participation and patient-centered outcomes are improved compared to the more common standardized approaches they tend to use now.

In this study, the investigators will compare the effectiveness of patient-driven diabetes SMAs to standardized diabetes SMAs. The curriculum to be used is Targeted Training for Illness Management (TTIM), a 6-session modular group intervention for chronic illness self-management, and has been tested in diabetes. The standardized group visit model will consist of diabetes SMAs with the full TTIM 6-session curriculum, led by a health educator. For the patient-driven SMAs, patients choose the topics and the order of sessions from the TTIM curriculum, which is delivered collaboratively by the multidisciplinary care team consisting of several professional providers (health educator, medical provider, and behavioral health provider) and a lay worker (diabetes peer mentor). The primary patient-centered outcome, selected by patient stakeholders, is diabetes distress. Secondary outcomes include autonomy support and diabetes self-management behaviors, clinical outcomes (hemoglobin A1c, blood pressure, and body mass index), patient reach and engagement, and practice-level value and sustainability. Patient, caregiver, practice, health plans, and research stakeholders will be engaged in all aspects of the research. Patients and other stakeholders will inform the process of implementation of patient-driven and standardized SMAs, help finalize the research protocol (including data collection and recruitment), and contribute to interpretation of findings and dissemination of findings, including messages that help other patients make decisions about whether or not to participate in SMAs.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be:

  1. at least 18 years old,
  2. have Type II Diabetes, and
  3. receive care in a participating practice.
* For a practice to be eligible, they must be;

  1. a Federally Qualified Health Center,
  2. a private primary care practice, or
  3. Community Mental Health Center with primary care,
  4. They need to have

     1. a current panel of at least 150 adult patients with Type 2 Diabetes, and
     2. access to health educators, Behavioral Health Professionals, and diabetes peer mentors.

Exclusion Criteria:

* Are currently pregnant or plan to become pregnant in the next six months,
* Have limited cognitive ability due to dementia or a developmental disorder,
* Less than one year of life expectancy, or
* Plan to leave the area in the next year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1085 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Kwan, PHD, MSPH, Principal Investigator — University of Colorado, Denver; Jeanette Waxmonsky, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The Investigators will be sharing results in aggregate form via publications and reports to the funder.

REFERENCES:
- [Derived] Holtrop JS, Gurfinkel D, Nederveld A, Reedy J, Rubinson C, Kwan BM. What works in implementing shared medical appointments for patients with diabetes in primary care to enhance reach: a qualitative comparative analysis from the Invested in Diabetes study. Implement Sci Commun. 2024 Jul 24;5(1):82. doi: 10.1186/s43058-024-00608-6. PMID 39049078
- [Derived] Kwan BM, Dickinson LM, Dailey-Vail J, Glasgow RE, Gritz RM, Gurfinkel D, Hester CM, Holtrop JS, Hosokawa P, Lanigan A, Nease DE Jr, Nederveld A, Phimphasone-Brady P, Ritchie ND, Sajatovic M, Wearner R, Begum A, Carter M, Carrigan T, Clay B, Downey D, Koren R, Trujillo SA, Waxmonsky JA. Comparative Effectiveness of Patient-Driven versus Standardized Diabetes Shared Medical Appointments: A Pragmatic Cluster Randomized Trial. J Gen Intern Med. 2024 Nov;39(15):2970-2979. doi: 10.1007/s11606-024-08868-7. Epub 2024 Jun 28. PMID 38943014
- [Derived] Nederveld A, Phimphasone-Brady P, Gurfinkel D, Waxmonsky JA, Kwan BM, Holtrop JS. Delivering diabetes shared medical appointments in primary care: early and mid-program adaptations and implications for successful implementation. BMC Prim Care. 2023 Feb 17;24(1):52. doi: 10.1186/s12875-023-02006-8. PMID 36803773
- [Derived] Holtrop JS, Gurfinkel D, Nederveld A, Phimphasone-Brady P, Hosokawa P, Rubinson C, Waxmonsky JA, Kwan BM. Methods for capturing and analyzing adaptations: implications for implementation research. Implement Sci. 2022 Jul 29;17(1):51. doi: 10.1186/s13012-022-01218-3. PMID 35906602
- [Derived] Glasgow RE, Gurfinkel D, Waxmonsky J, Rementer J, Ritchie ND, Dailey-Vail J, Hosokawa P, Dickinson LM, Kwan BM. Protocol refinement for a diabetes pragmatic trial using the PRECIS-2 framework. BMC Health Serv Res. 2021 Oct 2;21(1):1039. doi: 10.1186/s12913-021-07084-x. PMID 34598702
- [Derived] Dickinson LM, Hosokawa P, Waxmonsky JA, Kwan BM. The problem of imbalance in cluster randomized trials and the benefits of covariate constrained randomization. Fam Pract. 2021 Jun 17;38(3):368-371. doi: 10.1093/fampra/cmab007. No abstract available. PMID 33677530
- [Derived] Kwan BM, Dickinson LM, Glasgow RE, Sajatovic M, Gritz M, Holtrop JS, Nease DE Jr, Ritchie N, Nederveld A, Gurfinkel D, Waxmonsky JA. The Invested in Diabetes Study Protocol: a cluster randomized pragmatic trial comparing standardized and patient-driven diabetes shared medical appointments. Trials. 2020 Jan 10;21(1):65. doi: 10.1186/s13063-019-3938-7. PMID 31924249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited into shared medical appointments as part of their usual care for type 2 diabetes by participating practices from January 4, 2019 to September 30, 2021.
Pre-assignment Details: Randomization occurred at the practice level via Covariate Constrained Randomization. Patients seeking treatment in a practice assigned to the Standardized or the Patient-Driven condition received that treatment condition. Patients who were deemed ineligible for the study because they had type 1 diabetes or were pregnant during the study were removed from the analysis.
Period: Overall Study
Arm/Group | Standardized SMA | Patient-driven SMA
Started (Practices were allowed to begin cohorts of shared medical appointments at any time during the recruitment window (1/4/2019-9/30/2021).) | 576 | 509
Completed (Patients completed shared medical appointments at any time during the study implementation window (1/4/2019-12/31/2021).) | 558 | 504
Not Completed | 18 | 5
Not completed — Protocol Violation | 4 | 3
Not completed — No session data recorded | 14 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standardized SMA | Patient-driven SMA | Total
Number analyzed (Participants) | 558 | 504 | 1062
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (11.2) | 61.0 (11.6) | 60.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347 | 278 | 625
  Male | 211 | 226 | 437
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 137 | 155 | 292
  Not Hispanic or Latino | 414 | 319 | 733
  Unknown or Not Reported | 7 | 30 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 63 | 3 | 66
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 51 | 80
  White | 433 | 353 | 786
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 29 | 93 | 122
Diabetes Distress Scores [Mean (Standard Deviation); unit: units on a scale] — Diabetes Distress Scale (DDS-17) measures the worries, concerns and fears among individuals with diabetes over time as they struggle with managing diabetes. The DDS is a 17-item self-report instrument. Each of the 17 items is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem." The scale yields an overall distress score based on the average responses for all items. Average score of < 2.0 = reflects little or no distress; between 2.0 and 2.9 = reflects moderate distress; > 3.0 = reflects high distress. A total score of >2.0 is considered clinically significant.
  units on a scale | 2.2 (0.9) | 2.1 (1.0) | 2.2 (0.9)
Hemoglobin A1c [Mean (Standard Deviation); unit: % of hemoglobin coated in glucose] | 8.3 (2.0) | 8.3 (2.1) | 8.3 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Distress - Change in Patient Reported Outcomes (PROs)
Description: Comparison of change in patient-reported outcomes around diabetes distress for patients in either SMA group. Measured by the Diabetes Distress Scale (DDS-17). The DDS-17 measures the worries, concerns and fears among individuals with diabetes over time as they struggle with managing diabetes. The DDS is a 17-item self-report instrument. Each of the 17 items is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem." The scale yields an overall distress score based on the average responses for all items.
  Average score of < 2.0 = reflects little or no distress Average score between 2.0 and 2.9 = reflects moderate distress Average score > 3.0 = reflects high distress A total score > 2.0 (moderate distress) is considered clinically significant
Time Frame: At end of 6 group visits (time differs by practice, up to 6 months)
Population: Patients receiving SMAs as part of standard care at practices randomized to delivering either the Standardized or Patient-Driven model
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standardized SMA | Patient-driven SMA
Number analyzed (Participants) | 558 | 504
score on a scale | 1.9 (0.8) | 1.9 (0.8)
Statistical Analysis 1: Comparison: Standardized SMA vs Patient-driven SMA; We hypothesized that patients in Patient-Driven SMAs would have greater reductions in Diabetes Distress than those in Standardized SMAs. We expected seeing an effect size of a .6 unit decrease (.30) in Standardized SMAs and 1.2 unit decrease (.60) in Patient-Driven SMAs. We estimate we have >80% power to detect effect sizes between .29 (ICC=3%) and .34 (ICC=5%); Test type: Superiority; p = 0.04, Mixed Models Analysis — Linear Mixed Model adjusted for a priori patient covariates: Race/Ethnicity, Gender, Health Literacy, Food Availability, Charlson Score, Mental Illness, Substance use. Adjusted P-value represents the significance test for the time x group interaction

2. Secondary Outcome: Change in Patient HbA1c
Description: Comparison of change in patient HbA1c levels for patients in either SMA group. Measured by Electronic Medical Record data. It evaluates the average amount of glucose in the blood by measuring the percentage of glycated (glycosylated) hemoglobin
Time Frame: At end of 6 group visits (time differs by practice, up to 6 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %HbA1c
Arm/Group | Standardized SMA | Patient-driven SMA
Number analyzed (Participants) | 558 | 504
%HbA1c | 7.8 (1.9) | 7.9 (1.8)
Statistical Analysis 1: Comparison: Standardized SMA vs Patient-driven SMA; We hypothesized that patients in the Patient-Driven condition would have a greater reduction in HbA1c than patients in the Standardized condition. We estimate we have >80% power to detect effect sizes between .29 (ICC=3%) and .34 (ICC=5%); Test type: Superiority; p = 0.82, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: N/A - not monitored or collected
Description: There were no adverse health conditions collected as patients were receiving 2 versions of usual care and the intervention did not collect additional data on patients. "All-Cause Mortality", "Serious Adverse Events", and "Other (non-serious AEs) were not monitored/assessed.
Arm/Group | Standardized SMA | Patient-driven SMA
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT03590041/Prot_SAP_001.pdf
  • Informed Consent Form (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT03590041/ICF_000.pdf